CLINICAL TRIAL: NCT03124420
Title: Intraluminal Therapy for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tai-cherng Liou, MD, Clinical associate professor, Department of Medicine, Mackay Medical College, New Taipei City, Taiwan, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17MMHIS020
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Infection; Eradication therapy; Antibiotics
MeSH Terms: conditions — Helicobacter Infections | interventions — Lansoprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Intervention Model Description: Group A: 7-day triple therapy for patients fail to achieve intraluminal eradication Group B: 14-day triple therapy for patients fail to achieve intraluminal eradication
Who Masked: Investigator
Masking Description: open labeled, randomized control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Drug: 7-day triple therapy) (Active Comparator): Intervention : Drug: 7-day triple therapy. Patients fail to achieve intraluminal eradication of H. pylori will be randomly assigned to the oral antibiotics rescue therapies with standard 7-day triple therapy ( lansoprazole 30 mg b.i.d., amoxicillin 1 g b.i.d. and clarithromycin 500 mg b.i.d. for 7 days)
  Interventions: Drug: Lansoprazole; Drug: Amoxicillin; Drug: Clarithromycin
- Group B (Drug: 14-day triple therapy) (Sham Comparator): Intervention : Drug: 14-day triple therapy. Patients fail to achieve intraluminal eradication of H. pylori will be randomly assigned to the oral antibiotics rescue therapies with standard 14-day triple therapy ( lansoprazole 30 mg b.i.d., amoxicillin 1 g b.i.d. and clarithromycin 500 mg b.i.d. for 14 days).
  Interventions: Drug: Lansoprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Lansoprazole — Group A: lansoprazole 30 mg b.i.d. for 7 days Group B: lansoprazole 30 mg b.i.d. for 14 days
  Other Names: Takepron
Drug: Amoxicillin — Group A: amoxicillin 1 g b.i.d. for 7 days Group B: amoxicillin 1 g b.i.d. for 14 days
  Other Names: Supercillin
Drug: Clarithromycin — Group A: clarithromycin 500 mg b.i.d. for 7 days Group B: clarithromycin 500 mg b.i.d. for 14 days
  Other Names: Klaricid

SUMMARY:
Helicobacter pylori (H. pylori) is the most common chronic bacterial infection in humans.

The prevalence of H. pylori is about 30~50% in the Western adult population. It is estimated that about 50% of people are infected with this bacterium in Taiwan. Many studies have shown that H. pylori is an important causal factor of chronic gastritis, peptic ulcer disease, gastric cancer and gastric lymphoma. The World Health Organization classified H. pylori as a Group 1 carcinogen in 1994. Endoscopic examination is indicated to confirm the above diagnosis for patient with H. pylori infection. Eradication of H. pylori infection reduces the risk of gastric cancer and recurrence of peptic ulcer disease. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. Several strategies have been proposed to overcome the declining eradication rate, including (1) extending the treatment duration of triple therapy to 14 days; (2) the use of bismuth quadruple therapy which contains bismuth, a proton pump inhibitor, and two antibiotics (usually metronidazole and tetracycline); (3) non-bismuth quadruple therapy (concomitant therapy) which contains a proton pump inhibitor and three antibiotics (usually amoxicillin, metronidazole, and clarithromycin); (4) sequential therapy which contains a proton pump inhibitor (PPI) plus amoxicillin for five days, followed by a PPI plus clarithromycin and tinidazole for another five days. The investigators aim to improve the eradication rate of H. pylori infection while an endoscopic examination is performed.

DETAILED DESCRIPTION:
During the endoscopic examination, patient is sedated with intravenous Dormicum 5mg (5mg/1ml/amp), the vital signs will be closely monitored by physiological monitor (PHILIPS SureSigns VM6). The treatment will be terminated immediately if unstable vital sign detected or if patient asks for termination. With endoscope apparatus, the gastric mucous is irrigated with acetylcysteine solution and the pH value of gastric juice will be measured with the pH test strips before irrigation and after irrigation. The investigators dispense medicaments containing three kinds of antibiotics powder (Amoxicillin 3 gm、Metronidazole 2 gm and Clarithromycin 1 gm) on the surface of gastric mucosa and duodenal mucosa of duodenal bulb as evenly as possible. After the intraluminal therapy, patients will rest for 30 to 60 minutes and go home if the effect of sedation subsided. Patients can take meal if no abdominal discomfort. Patients will receive tests for serum Helicobacter pylori immunoglobulin G, liver function and renal function 3 to 7 days after the intraluminal therapy. C13-Urea breath test (UBT) will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy. Stool H. pylori Antigen will be used to assess the short term recurrence of H. pylori 4-6 months after successful intraluminal therapy . Patients fail to achieve intraluminal eradication of H. pylori will be randomly assigned to the oral antibiotics rescue therapies with standard triple therapy for either 7 days (Group A) or 14 days (Group B). C13-UBT will be used to assess the existence of H. pylori 6 weeks after the rescue triple therapy. Overall eradication rates after the first line intraluminal therapy and the oral antibiotics rescue therapies will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged greater than 20 years and less than 75 years
2. Patients have H. pylori infection without prior eradication therapy
3. Patients are willing to receive the intraluminal therapy. The written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

1. Children and teenagers aged less than 20 years, and adult greater than 75 years
2. Contraindication for endoscopic examination or food retention in the gastric lumen.
3. History of gastrectomy; Gastroduodenal stenosis、deformity or obstruction; Gastroduodenal malignancy, including adenocarcinoma and lymphoma
4. Contraindication to treatment drugs: previous allergic reaction to antibiotics (amoxicillin, clarithromycin, metronidazole), Proton pump inhibitors (lansoprazole), Acetylcystein and Sucralfate; pregnant or lactating women
5. Severe concurrent acute or chronic illness: renal failure, cirrhosis of liver, incurable malignant disease
6. Patients who cannot give informed consent by himself or herself.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Eradication rate in the intraluminal therapy | 6 weeks after finishing therapy
  C13-UBT will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy

SECONDARY OUTCOMES:
Eradication rates in the two groups of rescue oral antibiotics therapies. | 6 weeks after finishing therapy
  C13-UBT will be used to assess the existence of H. pylori 6 weeks after finishing rescue oral antibiotics therapies.
Overall eradication rates | 3-6 months after finishing intraluminal therapy
  Overall eradication rates after the first line intraluminal therapy and the oral antibiotics rescue therapies. Overall eradication rates after the first line intraluminal therapy and the oral antibiotics rescuOverall eradication rates after the first line intraluminal therapy and the oral antibiotics rescue therapies. e therapies.
Short term recurrent rate | 3-6 months after intraluminal therapy.
  To assess the short term recurrent rate 3-6 months after successful intraluminal therapy.
  Stool H. Pylori Ag will be used to assess the short term recurrence of H. pylori 3-6 months after successful intraluminal therapy .
Incidence of adverse effects in the intraluminal therapy. | within 7 days after finishing the intraluminal therapy
  Incidence of adverse effects were evaluated for Participants who had or had not finished the intraluminal therapy

OTHER OUTCOMES:
Evaluate eradication outcome of intraluminal therapy | 6 weeks after finishing therapy
  Evaluate eradication outcome by endoscopy urease test, the pH value of gastric juice or urea breath test

CONTACTS AND LOCATIONS:
Overall Officials: Tai-cherng Liou, MD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YC, Chen YP, Ho CY, Liu TW, Chu CH, Wang HY, Liou TC. The Impact of Gastric Juice pH on the Intraluminal Therapy for Helicobacter pylori Infection. J Clin Med. 2020 Jun 14;9(6):1852. doi: 10.3390/jcm9061852. PMID 32545856
- [Derived] Liou TC, Liao PH, Lin YC, Chu CH, Shih SC. Intraluminal therapy for Helicobacter pylori infection. J Gastroenterol Hepatol. 2019 Aug;34(8):1337-1343. doi: 10.1111/jgh.14627. Epub 2019 Feb 25. PMID 30734357